CLINICAL TRIAL: NCT01714843
Title: Phase II Study of ASP0456 - A Double-blind, Placebo-controlled, Parallel-group, Comparative Study in Patients With Constipation-predominant Irritable Bowel Syndrome
Brief Title: A Study to Evaluate the Effect of ASP0456 in Patients With Constipation Predominant Irritable Bowel Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0456-CL-0021
Record Dates: First submitted 2012-10-22; First posted 2012-10-26 (Estimated); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Constipation-predominant Irritable Bowel Syndrome (IBS-C)
Keywords: irritable bowel syndrome (IBS); linaclotide; constipation; ASP0456
MeSH Terms: conditions — Irritable Bowel Syndrome; Constipation | interventions — linaclotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- ASP0456 lowest dose group (Experimental): oral
  Interventions: Drug: linaclotide
- ASP0456 low dose group (Experimental): oral
  Interventions: Drug: linaclotide
- ASP0456 middle dose group (Experimental): oral
  Interventions: Drug: linaclotide
- ASP0456 high dose group (Experimental): oral
  Interventions: Drug: linaclotide
- placebo group (Placebo Comparator): oral
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: linaclotide — oral
  Other Names: ASP0456
  Arms: ASP0456 high dose group; ASP0456 low dose group; ASP0456 lowest dose group; ASP0456 middle dose group
Drug: placebo — oral
  Arms: placebo group

SUMMARY:
This study is to investigate the efficacy, safety, and plasma concentration change of ASP0456 in patients with constipation-predominant irritable bowel syndrome.

DETAILED DESCRIPTION:
This study is a multicenter, double-blind, placebo-controlled, parallel-group, comparative study to investigate dose-responses of efficacy, safety, and pharmacokinetics of ASP0456 in patients with constipation-predominant irritable bowel syndrome (IBS-C) according to the Rome III Diagnostic Criteria (2006 revised edition, established by the Rome III Committee) after oral administration of ASP0456.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had abdominal pain or discomfort repeatedly for at least 3 days per month during the 3 months before screening examination associated with at least 2 out of the following 3 conditions: (1) Improvement with defecation; (2) Onset associated with a change in frequency of stool; and (3) Onset associated with a change in form (appearance) of stool, and had the above symptom (IBS symptom) 6 months or more before the screening examination period.
* Patients with ≥25% of stools hard or lumpy (with each bowel movement occurring without antidiarrheal, laxative, suppository or enema) and <25% of them loose (mushy) or watery during the 3 months before the screening examination.
* Patients who had pancolonoscopy or contrast enema (or sigmoidoscopy) after the onset of IBS symptom and had no organic changes.

Exclusion Criteria:

* Patients with a history of surgical resection of the stomach, gallbladder, small intestine or large intestine
* Patients with other concurrent diseases that may affect the digestive tract passage or large intestinal function
* Patients with other concurrent diseases that may affect the assessment of abdominal pain/discomfort
* Patients with blood pressure, pulse rate, clinical laboratory test, or 12-lead ECG at the time of screening examination that was rated as Grade 2 or greater on the "Severity Criteria for Drug Adverse Reaction" and judged to be clinically significant

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 559 (Actual)
Dates: Start 2012-08-10 (Actual); Primary Completion 2013-12-07 (Actual); Study Completion 2013-12-07 (Actual)

PRIMARY OUTCOMES:
Global assessment of relief of IBS symptoms Responder | Weekly for 12 weeks

SECONDARY OUTCOMES:
SBM (Spontaneous Bowel Movement) Responder | Weekly for 12 weeks
CSBM (Complete SBM) Responder | Weekly for 12 weeks
Abnormal bowel habits improvement Responder | Weekly for 12 weeks
Abdominal pain/discomfort relief Responder | Weekly for 12 weeks
Changes in weekly average of SBM frequency | Weekly for 12 weeks
Changes in weekly average of CSBM frequency | Weekly for 12 weeks
Changes in weekly average of stool form scores | Weekly for 12 weeks
Changes in weekly average of abdominal pain/discomfort severity | Weekly for 12 weeks
Changes in weekly average of straining severity | Weekly for 12 weeks
Changes in IBS-QOL-J scores (entire scores or scores on the sub-scales) | Weekly for 12 weeks
Safety assessed by the incidence of adverse events, vital signs, clinical laboratory tests and 12-lead ECGs | for 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (4):
- Japan (4):
  - Hokkaido
  - Kansai
  - Kantou
  - Kyusyu

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=206